CLINICAL TRIAL: NCT04590131
Title: Efficacy and Safety Comparison of the Endovascular (Recanalization With Angioplasty and Stenting With Biomimetic Interwoven Nitinol Stent) and the Hybrid (Recanalization With Angioplasty and Stenting With Biomimetic Interwoven Nitinol Stent, Supplemented With Fasciotomy in Hunter's Canal) Surgical Methods for the Treatment of Prolonged Atherosclerotic Lesions of the Femoral-popliteal Segment Above the Knee, TASC II, Type D
Brief Title: Efficacy and Safety Comparison of the Endovascular and the Hybrid Methods for the Treatment of Prolonged Atherosclerotic Lesions of the Femoral-popliteal Segment Above the Knee, TASC II, Type D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sosudi3
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Atherosclerosis; Ischemia Limb; Superficial Femoral Artery Occlusion; Popliteal Artery Occlusion; Stent Complication
Keywords: interwoven nitinol stent; atherosclerosis; prolonged occlusion of SFA; endovascular treatment; hybrid revascularization; TASC II, type D
MeSH Terms: conditions — Atherosclerosis | interventions — Angioplasty; Stents

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, open-label, pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hubrid revaskularization (Experimental): Patients (n=50) with recanalization of the femoral-popliteal arterial segment above the knee with angioplasty and stenting with a biomimetic interwoven nitinol stent, supplemented by fasciotomy in Hunter's canal.
  Interventions: Procedure: recanalization of the femoral-popliteal arterial segment above the knee with angioplasty and stenting with a biomimetic interwoven nitinol stent, supplemented by fasciotomy in Hunter's canal.
- Endovascular treatment (Active Comparator): Patients (n=50) with recanalization of the femoral-popliteal arterial segment above the knee with angioplasty and stenting with a biomimetic interwoven nitinol stent.
  Interventions: Procedure: recanalization of the femoral-popliteal arterial segment above the knee with angioplasty and stenting with a biomimetic interwoven nitinol stent.

INTERVENTIONS:
Procedure: recanalization of the femoral-popliteal arterial segment above the knee with angioplasty and stenting with a biomimetic interwoven nitinol stent, supplemented by fasciotomy in Hunter's canal. — Under local anesthesia, a standard endovascular approach is performed. Transluminal or subintimal recanalization of the occluded arterial segment is performed with a hydrophilic guidewire. Next, balloon angioplasty of the recanalized segment is performed. After control angiography, a biomimetic interwoven nitinol stent is placed throughout the lesion. Immediately after the stenting procedure, under local anesthesia, access to the distal part of the SFA at the outlet of Hunter's canal and 1 portion of the popliteal artery is performed. The lamina vastoadductoria is dissected. The wound is sutured in layers. An aseptic bandage is applied. Drug therapy includes pre-procedure clopidogrel (160-300 mg/day), starting at least one day before, and intra-procedure heparin (100 U / kg body weight intravenously). After the procedure, all patients have prescribed double antiplatelet therapy (aspirin+clopidogrel (75 mg per day) within 6 months and then aspirin 75 mg for a long time.
  Arms: Hubrid revaskularization
Procedure: recanalization of the femoral-popliteal arterial segment above the knee with angioplasty and stenting with a biomimetic interwoven nitinol stent. — Under local anesthesia, a standard endovascular approach is performed and the affected arterial segment is visualized. Transluminal or subintimal recanalization of the occluded arterial segment is performed with a hydrophilic guidewire. Next, balloon angioplasty of the recanalized segment is performed. After control angiography, a biomimetic interwoven nitinol stent is placed throughout the lesion. Drug therapy includes pre-procedure clopidogrel (160-300 mg/day), starting at least one day before, and intra-procedure heparin (100 U / kg body weight intravenously). After the procedure, all patients have prescribed double antiplatelet therapy (aspirin+clopidogrel (75 mg per day) within 6 months and then aspirin 75 mg for a long time.
  Arms: Endovascular treatment

SUMMARY:
A recent study, where the authors studied the effectiveness of stenting of prolonged lesions (>200 mm) of the femoral-popliteal segment with nitinol stents (TASC II, D), showed unsatisfactory primary patency rates (45%) within 2 years follow up (Lin et al, 2015). One of the possible solutions to the problem of breakage of stents in the femoral-popliteal position is a modified method of their manufacture by braiding from nitinol wire. Another possible solution to the problem of stent breakage in the femoral-popliteal position is fasciotomy in Gunter's canal with dissection of the lamina vasto-adductoria. According to a pilot randomized study (Karpenko et al, 2019), the primary patency at 24 months was 60% in the stenting group supplemented with fasciotomy in Gunter's canal, and 28.5% in the stenting group without fasciotomy. These facts prove the need for a comparative study on a cohort of patients using a biomimetic interwoven nitinol stent. This is a pilot prospective, randomized, open-label study. The main objective of the study is to compare the clinical efficacy and safety of two methods of treating prolonged atherosclerotic lesions (TASC II, type D) of the arteries of the femoropopliteal segment above the knee.

DETAILED DESCRIPTION:
A recent study, where the authors studied the effectiveness of stenting of prolonged lesions (>200 mm) of the femoral-popliteal segment with nitinol stents (TASC II, D), showed unsatisfactory primary patency rates (45%) within 2 years follow up (Lin et al, 2015). One of the possible solutions to the problem of breakage of stents in the femoral-popliteal position is a modified method of their manufacture by braiding from nitinol wire. Another possible solution to the problem of stent breakage in the femoral-popliteal position is fasciotomy in Gunter's canal with dissection of the lamina vasto-adductoria. According to a pilot randomized study (Karpenko et al, 2019), the primary patency at 24 months was 60% in the stenting group supplemented with fasciotomy in Gunter's canal, and 28.5% in the stenting group without fasciotomy. These facts prove the need for a comparative study on a cohort of patients using a biomimetic interwoven nitinol stent. This is a pilot prospective, randomized, open-label study. The main objective of the study is to compare the clinical efficacy and safety of two methods of treating prolonged atherosclerotic lesions (TASC II, type D) of the arteries of the femoropopliteal segment above the knee.

Screening It is performed in patients with a verified diagnosed occlusive lesion of the femoropopliteal segment above the knee (type D by TASC II classification), with chronic limb ischemia (3-6 categories by Rutherford classification). Assessment of inclusion / exclusion criteria, assigning a patient number.

Study inclusion Collecting baseline information about the patient (anamnesis, including information about concomitant therapy, data from the initial physical examination, ultrasound data of the lower limb arteries, CT-angiography data, assessment of the quality of life using the SF-36 questionnaire). Randomization using the envelope method to one group or another.

Surgical intervention:

Group 1 (n=50): Recanalization of prolonged occlusion of the arteries of the femoral-popliteal segment above the knee with angioplasty and stenting with a biomimetic interwoven nitinol stent; Group 2 (n=50): Recanalization of prolonged occlusion of the arteries of the femoropopliteal segment above the knee with angioplasty and stenting with a biomimetic interwoven nitinol stent, supplemented by fasciotomy in Gunter's canal.

Follow up: 6, 12, 24 months.

Performed:

Triplex ultrasound of one lower limb (restenosis, thrombosis, stent breakage); Radiography of the operated limb in two projections, for patients in whom a stent breakage is suspected according to ultrasound; Consultation with a cardiovascular surgeon. For each patient participating in the study, a CRF is filled out in a form convenient for the Investigator. The creation of a folder "Investigator's file" is provided, which stores all the necessary documents provided for by the rules of "Good Clinical Practice".

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years;
* CLI category 3 - 6 by Rutherford classification;
* Prolonged atherosclerotic occlusive lesion of the femoropopliteal arterial segment above the knee (Type D by TASC II classification), confirmed by CT or arteriography;
* De novo lesion;
* Patient informed consent.

Exclusion Criteria:

* Age < 18;
* Potentially pregnant women;
* Asymptomatic lesion;
* Acute ischemia;
* Previous treatment on the affected segment;
* Not atherosclerotic lesion;
* Severe comorbidity with a life expectancy of fewer than 2 years;
* Contraindications to antiplatelet therapy;
* Patient participation in another clinical trial;
* Inability to monitor the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 24 months
  primary patency was defined as absence of occlusion or flow-limiting stenosis (peak systolic velocity [PSV] ratio >2.5) of the treated segment including 1 cm proximal and distal of the anastomosis;
primary assisted patency | 24 months
  primary assisted patency was defined as a secondary procedure is performed to prevent failure (i.e., in a flow-limiting stenosis [PSV ratio >2.5] in a still-patent segment of stent or bypass, including the anastomoses;
secondary patency | 24 months
  secondary patency was defined as a secondary procedure performed for graft or stent occlusion in an afterward patent vessel;

SECONDARY OUTCOMES:
MALE | 24 months
  major adverce limb events
Safety of the methods in the early postoperative period | 30 days
  hematoma of the surgical access area, peripheral neuropathy, purulent-infectious complications of the surgical access area
MACE | 24 months
  major adverce cardio-vascular events
Assessment of the quality of life in patients after surgical treatment | 24 months
  SF-36 questionary

CONTACTS AND LOCATIONS:
Locations (1):
- Meshalkin Research Institute of Pathology of Circulation, Novosibirsk, Novosibirsk Area, Russia

IPD SHARING:
Plan to Share IPD: No